CLINICAL TRIAL: NCT05077254
Title: A Randomized Study to Evaluate Antibody Response to an Additional Dose of SARS-CoV-2 Vaccination With and Without Immunosuppression Reduction in Kidney and Liver Transplant Recipients
Brief Title: COVID Protection After Transplant-Immunosuppression Reduction
Acronym: CPAT-ISR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: PPD Development, LP (Industry); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT COVID19-TB-03; U01AI138897 (NIH); NIAID CRMS ID#: 38892 (Other: DAIT NIAID)
Record Dates: First submitted 2021-10-12; First posted 2021-10-14 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Kidney Transplant Recipients; Liver Transplant Recipients
Keywords: mRNA COVID-19 vaccines; SARS-CoV-2 antibody response; immunosuppression (IS); coronavirus infectious disease 19; COVID-19; severe acute respiratory syndrome coronavirus type 2; SARS-CoV-2 protection
MeSH Terms: conditions — COVID-19 | interventions — CVnCoV COVID-19 vaccine; BNT162 Vaccine; 2019-nCoV Vaccine mRNA-1273; COVID-19 Vaccines; Immunosuppression Therapy; Mycophenolic Acid; Tacrolimus; Standard of Care

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to:
  * A study dose of mRNA COVID-19 vaccine only, or
  * Immunosuppression (IS) reduction plus a study dose of mRNA COVID-19 vaccine. IS reduction will be based on the participant's IS regimen upon study entry, in accordance with the study's protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Pfizer-BioNTech COVID-19 Vaccine 2023-2024 + SOC IS Regimen (Experimental): Participants will receive a study dose (1 dose) of the Pfizer-BioNTech COVID-19 Vaccine 2023-2024 and will continue to take their standard of care transplant immunosuppressive medications without alterations in schedule and dosing.
  SOC IS: Standard of Care transplant immunosuppression regimen
  Interventions: Biological: Pfizer-BioNTech COVID-19 Vaccine 2023-2024; Drug: SOC IS Regimen
- Pfizer-BioNTech COVID-19 Vaccine 2023-2024 + SOC IS Reduction (Experimental): Participants will receive an additional dose (1 dose) of the Pfizer-BioNTech COVID-19 Vaccine 2023-2024, with concurrent reduction of their standard of care transplant immunosuppression regimen (IS), per protocol.
  SOC IS Reduction: Standard of Care transplant immunosuppression regimen reduction, per protocol
  Interventions: Biological: Pfizer-BioNTech COVID-19 Vaccine 2023-2024; Drug: SOC IS Reduction
- Moderna COVID-19 Vaccine 2023-2024 + SOC IS Regimen (Experimental): Participants will receive an additional dose (1 dose) of the Moderna COVID-19 Vaccine 2023-2024 and will continue to take their standard of care transplant immunosuppressive medications without alterations in schedule and dosing.
  SOC IS: Standard of Care transplant immunosuppression regimen
  Interventions: Biological: Moderna COVID-19 Vaccine 2023-2024; Drug: SOC IS Regimen
- Moderna COVID-19 Vaccine 2023-2024 + SOC IS Reduction (Experimental): Participants will receive a study dose (1 dose) of the Moderna COVID-19 Vaccine 2023-2024, with concurrent reduction of their standard of care transplant immunosuppression regimen (IS), per protocol.
  SOC IS Reduction: Standard of Care transplant immunosuppression regimen reduction, per protocol
  Interventions: Biological: Moderna COVID-19 Vaccine 2023-2024; Drug: SOC IS Reduction

INTERVENTIONS:
Biological: Pfizer-BioNTech COVID-19 Vaccine 2023-2024 — Administration: One dose administered intramuscularly.
  Other Names: mRNA COVID-19 vaccine; BNT162b2 mRNA COVID-19 vaccine; SARS-CoV-2 RNA vaccine; Comirnaty
  Arms: Pfizer-BioNTech COVID-19 Vaccine 2023-2024 + SOC IS Reduction; Pfizer-BioNTech COVID-19 Vaccine 2023-2024 + SOC IS Regimen
Biological: Moderna COVID-19 Vaccine 2023-2024 — Administration: One dose administered intramuscularly.
  Other Names: mRNA COVID-19 vaccine; Moderna COVID-19 vaccine; SARS-CoV-2 vaccine; Spikevax
  Arms: Moderna COVID-19 Vaccine 2023-2024 + SOC IS Reduction; Moderna COVID-19 Vaccine 2023-2024 + SOC IS Regimen
Drug: SOC IS Regimen — Participants will continue to take their prescribed immunosuppression (IS) medications without alterations in schedule and dosing, per protocol instruction.
  Other Names: Standard of Care transplant immunosuppression regimen; Immunosuppression (IS); mycophenolate mofetil (MMF) or equivalent; tacrolimus
  Arms: Moderna COVID-19 Vaccine 2023-2024 + SOC IS Regimen; Pfizer-BioNTech COVID-19 Vaccine 2023-2024 + SOC IS Regimen
Drug: SOC IS Reduction — Participants will reduce their standard of care immunosuppression medications (IS) before and after the COVID-19 vaccine booster (1 dose), per protocol instruction.
  Other Names: Standard of Care (SOC) transplant immunosuppression regimen; Immunosuppression (IS) Reduction; mycophenolate mofetil (MMF) or equivalent; tacrolimus
  Arms: Moderna COVID-19 Vaccine 2023-2024 + SOC IS Reduction; Pfizer-BioNTech COVID-19 Vaccine 2023-2024 + SOC IS Reduction

SUMMARY:
This study will enroll individuals who have:

* Completed primary series of mRNA COVID-19 vaccine, and
* An antibody response ≤ 2500 U/mL measured at least 30 days after the last dose of vaccine.

This group of patients is at high risk for severe COVID-19 disease due to pharmacologic immunosuppression and a high prevalence of non-transplant risk factors such as obesity and diabetes.

DETAILED DESCRIPTION:
This study is a randomized, open-label multi-site trial designed to induce an enhanced antibody response to severe acute respiratory syndrome coronavirus type 2 (SARS-CoV-2) in kidney and liver transplant recipients who have ≤ 2500 U/mL anti-spike antibody (as measured by the Roche Elecsys® anti-SARS-CoV-2 S assay) after a completed primary series (3 doses) of mRNA COVID-19 vaccines.

Participants will be randomized to either:

1. Receive a study dose of mRNA based COVID-19 vaccine (booster) with no change in their immunosuppressive regimen, or
2. Undergo a temporary, prescribed reduction in their maintenance immunosuppression (IS) regimen and receive a study dose (booster) of mRNA based COVID-19 vaccine.

Protocol Version 8.0 will include a booster dose of either Pfizer-BioNTech COVID-19 Vaccine 2023-2024 or Moderna COVID-19 Vaccine 2023-2024, with or without IS reduction.

Duration of study participation for interested and eligible individuals: 13 months.

ELIGIBILITY:
Inclusion Criteria:

Individuals who meet all the following criteria are eligible for enrollment as study participants-

1. Able to understand and provide informed consent
2. Individual ≥18 years of age.
3. Recipient of a kidney or liver transplant ≥12 months prior to enrollment, without allograft rejection in the 6 months preceding enrollment
4. Negative for anti-donor human leukocyte antigens (HLA) antibodies at screening (Central Lab Test Determination).
5. Currently taking one of the following tacrolimus-based immunosuppressive regimens:

   * Tacrolimus plus Mycophenolate Mofetil (MMF) or Mycophenolic Acid (MPA), with or without a corticosteroid
   * Tacrolimus with trough ≥ 5ng/mL with or without ≤5 mg of prednisone or equivalent
6. Received a minimum of 3 doses of either the Moderna coronavirus infectious disease 19 (COVID-19) vaccine or Pfizer-BioNTech COVID-19 vaccine
7. Participant must be ≥ 60 days after completion of primary vaccination or receipt of the most recent booster dose with any authorized or approved monovalent or bivalent COVID-19 vaccine at the time of study vaccine.
8. Serum antibody negative or low (titer ≤ 2500 U/mL) at ≥ 30 days from the last dose of mRNA COVID-19 vaccine and ≥ 30 days following receipt of a monoclonal antibody product or convalescent plasma for COVID-19, measured using the Roche Elecsys® anti-SARS-CoV-2 S assay.
9. Participant's transplant physician or midlevel practitioner who is clinically licensed to prescribe and manage immunosuppression must confirm the participant's eligibility based on medical history.

Exclusion Criteria:

Individuals who meet any of these criteria are not eligible for enrollment as study participants-

1. Currently on an immunosuppressive regimen different from the three regimens described in the Inclusion Criteria, for example (but not limited to) those including sirolimus, everolimus, belatacept, or azathioprine
2. Recipient of any allograft other than a kidney or liver
3. Participant is pregnant
4. Any past history of Donor Specific Antibody (DSA) using local site standards
5. Prior receipt of the Moderna COVID-19 Vaccine 2023-2024 or Pfizer-BioNTech COVID-19 Vaccine 2023-2024.
6. Currently taking any systemic immunosuppressive agent, other than their prescribed transplant immunosuppression
7. Known history of severe allergic reaction to any component of an authorized or licensed COVID-19 vaccine
8. Thrombotic events, myocarditis, or pericarditis temporally associated with a prior dose of COVID-19 vaccine
9. History of heparin-induced thrombocytopenia
10. Any change in transplant immunosuppression regimen (drug or dose) in response to suspected or proven rejection within the last 6 months
11. More than minimal graft dysfunction, in accordance with study definition
12. Receipt of any cellular depleting agent (e.g. antithymocyte globulins (ATG), rituximab, alemtuzumab, Cyclophosphamide) within 12 months preceding enrollment
13. Concurrent autoimmune disease at risk for exacerbation with immunosuppression reduction
14. Any untreated active infection including BK viremia >10^4 copies
15. Infection with human immunodeficiency virus (HIV)
16. Recent (within one year) or ongoing treatment for malignancy with the exception of:

    * Non- melanomatous skin cancer definitively treated by local therapy, and
    * Definitively treated carcinoma-in-situ of the cervix (Stage 0 cervical cancer)
17. Treatment or prophylaxis of COVID-19 with a monoclonal antibody product or convalescent plasma within 6 months preceding enrollment, or
18. Any past or current medical problems, treatments, or findings which, in the opinion of the investigator, may:

    * pose additional risks from participation in the study,
    * interfere with the candidate's ability to comply with study requirements, or
    * impact the quality or interpretation of the data obtained from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2025-02-21 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the -fold increase in antibody titer (using the Roche Elecsys® anti-SARS-CoV-2 S assay) from before receiving the study dose of vaccine to 30 days after the study dose of vaccine. | Day 30 After Study Vaccination
  Serum antibody titer will be measured using the Roche Elecsys®) severe acute respiratory syndrome coronavirus type 2 serological (anti-SARS-CoV-2) S assay.

SECONDARY OUTCOMES:
Frequency of Solicited Local Reactogenicity Adverse Events (AEs) to the mRNA-Based COVID-19 Vaccine | Through Day 7 Post Study Vaccination
  Safety measure after receipt of the study's COVID-19 mRNA vaccine.
Frequency of Solicited Local Allergic Reaction Adverse Events (AEs) to the mRNA-Based COVID-19 Vaccine | Through Day 7 Post Study Vaccination
  Safety measure after receipt of the study's COVID-19 mRNA vaccine.
Frequency of Solicited Systemic Reactogenicity Adverse Events (AEs) to the mRNA-Based COVID-19 Vaccine | Through Day 7 Post Study Vaccination
  Safety measure after receipt of the study's COVID-19 mRNA vaccine.
Frequency of Solicited Systemic Allergic Reaction Adverse Events (AEs) to the mRNA-Based COVID-19 Vaccine | Through Day 7 Post Study Vaccination
  Safety measure after receipt of the study's COVID-19 mRNA vaccine.
Frequency of Any Serious Adverse Events (SAEs) | Through Day 30 Post Study Vaccination
  Safety measure after receipt of the study's COVID-19 mRNA vaccine.
Frequency of Any Unsolicited Adverse Events (AEs) | Through Day 30 Post Study Vaccination
  Safety measure. An AE associated with the receipt of the study's COVID-19 mRNA vaccine and/or study mandated procedures.
Frequency of Any Serious Adverse Events (SAEs) | Through Day 60 Post Study Vaccination
  Safety measure after receipt of the study's COVID-19 mRNA vaccine.
Frequency of Any Serious Adverse Events (SAEs) | Through Day 365 Post Study Vaccination
  Safety measure after receipt of the study's COVID-19 mRNA vaccine.
Frequency of Any Unsolicited Adverse Events (AEs) | Through Day 365 Post Study Vaccination
  Safety measure. An AE associated with the receipt of of the study's COVID-19 mRNA vaccine and/or study mandated procedures.
Proportion of Participants Treated for Acute Cell-Mediated and/or Antibody-Mediated Allograft Rejection | Through Day 60 Post Study Vaccination
  Safety measure post receipt of the study's COVID-19 mRNA vaccine.
Proportion of Participants who Develop de Novo Donor-Specific Anti-Human Leukocyte Antigens (HLA) Antibody | Through Day 60 Post Study Vaccination
  Safety measure after receipt of the study's COVID-19 mRNA vaccine.
Proportion of Participants with Graft Loss | Through Day 60 Post Study Vaccination
  Safety measure after receipt of the study's COVID-19 mRNA vaccine.
Occurrence of Death Among Participants | Through Day 60 Post Study Vaccination
  Safety measure after receipt of the study's COVID-19 mRNA vaccine.
Frequency of Positive SARS-CoV-2 Test Results Using Real-Time Polymerase Chain Reaction (RT-PCR) | Baseline (Day 0, Prior to Study Vaccination), Month 1, 3, 6, 9 and 12
  A nasal mid-turbinate swab for SARS-CoV-2 PCR testing will be collected prior to administration of the COVID-19, at specified timepoints after receipt of vaccination and, in any case of suspected COVID-19 infection.
Occurrence of Symptomatic COVID-19 | Through Day 365 Post Study Vaccination
  Efficacy measure after receipt of the study's COVID-19 mRNA vaccine.
Occurrence of COVID-19 Requiring Hospitalization | Through Day 365 Post Study Vaccination
  Efficacy measure after receipt of the study's COVID-19 mRNA vaccine.
Change from Baseline in Anti-SARS-CoV-2 Antibody Levels at Day 30 | Baseline (Day 0, Prior to Study Vaccination),Day 30 After Study Vaccination
  Efficacy measure after receipt of the study's COVID-19 mRNA vaccine.
Change from Baseline in SARS-CoV-2 Antibody Levels | From Baseline (Day 0, Prior to Study Vaccination) to Day 365 Post Study Vaccination
  Efficacy measure after receipt of the study's COVID-19 mRNA vaccine.
Fold Increase in SARS-CoV-2 Antibody Levels: Limited to Participants With Detectable Antibody Levels at Baseline (Day 0) | Baseline (Day 0, Prior to Receipt of COVID-19 Study Vaccination), Day 30 After Study Vaccination
  Efficacy measure after receipt of the study's COVID-19 mRNA vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Dorry L. Segev, MD, PhD, Study Chair — Transplant Surgery, Johns Hopkins University School of Medicine; Peter S. Heeger, MD, Study Chair — Translational Transplant Research Center, Icahn School of Medicine at Mount Sinai; Christian P. Larsen, MD, DPhil, Study Chair — Emory Transplant Center, Emory University School of Medicine
Locations (15):
- United States (15):
  - University of California, San Diego, San Diego, California
  - University of California San Francisco Health, San Francisco, California
  - Emory Healthcare, Atlanta, Georgia
  - University of Illinois Health, Chicago, Illinois
  - Northwestern University, Evanston, Illinois
  - University of Iowa Hospitals, Iowa City, Iowa
  - Ochsner Health, New Orleans, Louisiana
  - Johns Hopkins Institute for Clinical and Translational Research: Broadway Adult Outpatient Clinical Research Unit, Baltimore, Maryland
  - NYU Langone Transplant Institute, New York, New York
  - Mt. Sinai Hospital, New York, New York
  - Weill Cornell Medicine, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Houston Methodist, Houston, Texas
  - University of Wisconsin-Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data upon completion of the study in: Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
Time Frame: On average, within 24 months after database lock for the trial.
Access Criteria: Open access.
URL: https://www.immport.org/home

REFERENCES:
- [Background] Werbel WA, Boyarsky BJ, Ou MT, Massie AB, Tobian AAR, Garonzik-Wang JM, Segev DL. Safety and Immunogenicity of a Third Dose of SARS-CoV-2 Vaccine in Solid Organ Transplant Recipients: A Case Series. Ann Intern Med. 2021 Sep;174(9):1330-1332. doi: 10.7326/L21-0282. Epub 2021 Jun 15. No abstract available. PMID 34125572
- See also: National Institute of Allergy and Infectious Diseases — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation — https://www.niaid.nih.gov/about/dait